CLINICAL TRIAL: NCT05541406
Title: Efficacy of a Multi-level School Intervention for LGBTQ Youth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH Funding Cuts
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Southern California (Other)
Responsible Party: Principal Investigator, Jeremy T. Goldbach, Masters & Johnson Distinguished Professor of Sexual Health and Education, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202208172; 1R01MD016082-01A1 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety; Post Traumatic Stress Disorder; Coping Behavior; Sexual Minority Stress; Suicidality; Substance Use; Bullying; Harassment
Keywords: LGBTQ+ Youth; LGBT Youth; Queer Youth
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Suicidal Ideation; Substance-Related Disorders; Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (Experimental): Schools will be assigned to either intervention or control schools. Students in intervention schools will receive the intervention in semester 1.
  Interventions: Behavioral: Proud & Empowered
- Control schools (Active Comparator): Students in control schools will receive no intervention
  Interventions: Behavioral: Proud & Empowered

INTERVENTIONS:
Behavioral: Proud & Empowered — Proud & Empowered! is a school-based intervention to decrease sexual minority stress and improve coping among LGBTQ students. It is administered by school counselors and trained social workers.

SUMMARY:
Efficacy of a Multi-level School Intervention for LGBTQ Youth

DETAILED DESCRIPTION:
The goal of this R01 grant is to test the efficacy of a theoretically informed, LGBTQ-affirming intervention (Proud & Empowered; P&E) alongside a school climate intervention (Make Space).

Sexual and gender minority adolescents (SGMA) experience victimization in schools at much higher rates than their peers, and although SGMA experience disparities in behavioral health outcomes compared to their heterosexual peers, interventions are scarce.

The investigators P&E intervention aims to allow youth participants to discuss their experiences of bullying and victimization, to build coping skills and to plan stress management strategies, while the investigators Make Space intervention is an indirect, environmental strategy aimed at improving overall school climate. The investigators goal will be achieved by completing three specific aims: 1) Determine participant-level efficacy of the intervention in an RCT with 24 schools (6-10 schools each year over 4 years); 2) Determine the school-wide intervention effects on (a) reporting of minority stress and behavioral health outcomes among all SGMA students and (b) perceptions of school climate (norms, attitudes, beliefs, bullying behaviors toward SGM youth, policies) among all students, and; 3) Examine factors that may affect intervention success (e.g., fidelity of implementation, barriers or facilitators to implementation, school or student characteristics) to prepare the intervention for future dissemination. This intervention has been tested in a previous, smaller, Feasibility study with 4 high schools.

ELIGIBILITY:
Inclusion Criteria:

* LGBTQ student in one of 24 high schools

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 228 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Sexual Minority Stress Inventory | Change between baseline and post-intervention/follow-up (12 weeks)
  54-item survey across 10 domains of minority stress. Assesses experiences of minority stress among adolescents. Each statement reflects past-30-day thoughts, feelings, and situations a person may have experienced, with response options of 1 = yes and 0 = no. A total score was calculated by summing the 54 items. The total score ranged from 0-54. Higher values correspond to a worse outcome, meaning the individual in question has had more stressful experiences.
Beck Anxiety Inventory (BAI) | Change between baseline and post-intervention/follow-up (12 weeks)
  21-item self-report assessment of anxiety symptoms. The total score is calculated by taking the sum of the 21 items. There are five responses an individual can choose from for each item, these being "Not at all" which is scored as a 1, "Mildly, but it didn't bother me much" which is scored as a 2, "Moderately -- It wasn't pleasant at times" which is scored as a 3, "Severely -- It bothered me a lot" which is scored as a 4, and "Decline to answer" which is scored as a 5. The total score ranges from 0-63. Higher values indicate higher self-reported anxiety: Score of 0-21 indicates low anxiety, Score of 22-35 indicates moderate anxiety, Scores of 36+ indicates potentially concerning levels of anxiety. Subscales are calculated through summation.
PTSD Checklist for DSM-5 (PCL-5) | Change between baseline and post-intervention/follow-up (12 weeks)
  20-item self-report assessment of post-traumatic stress disorder (PTSD) symptoms which addresses all 20 DSM-5 symptoms of PTSD. A total symptom severity score can be calculated by summing the scores for each of the 20 items. Each item has five possible responses including "Not at all" which is scored as a 0, "A little bit" which is scored as a 1, "Moderately" which is scored as 2, "Quite a bit" which is scored as a 3, and "Extremely" which is scored as a 4. The potential range of scores is 0-80. Higher scores indicate a worse outcome where the individual has higher severity of PTSD symptoms.
Beck Depression Inventory | Change between baseline and post-intervention/follow-up (12 weeks)
  21-item self-report assessment of depression symptoms and severity of depression. The items are rated on a 4-point scale ranging from 0-3 based on the severity of each item (e.g., 0=I do not feel sad, 1=I feel sad much of the time, 2=I am sad all the time, and 3=I am so sad or unhappy that I can't stand it). The total range of scores is from 0-63. Higher values indicate a worse outcome and indicates a greater severity of depression. Scores of 0-13 indicates minimal depression, scores of 14-19 indicates mild depression, scores of 20-28 indicates moderate depression, scores of 29-63 indicates severe depression. Subscale values are achieved through summation.
Coping Strategies Inventory | Change between baseline and post-intervention/follow-up (12 weeks)
  16-item assessment measuring specific coping strategies people use in response to stressful events. Individuals respond to 16 items, with each item assessing components of Problem Solving, Cognitive Restructuring, Social Support, Express Emotions, Problem Avoidance, Wishful Thinking, and Social Withdrawal. Individuals can respond in 5 different ways, these being "Never", "Seldom", "Sometimes", "Often", or "Almost Always". These responses are scored from 1-5 with "Never" being a 1 and "Almost Always" being a 5. The total score is a summation of item scores with a range from 16-80. Higher scores in a particular primary scale indicates that the individual implements that form of coping strategy more often.
Adapted CSSRS Suicide Questions (Columbia Suicide Severity Rating Scale) | Change between baseline and post-intervention/follow-up (12 weeks)
  Six items assessing current suicidality that were adapted from the longer, treatment-based Columbia Suicide Severity Rating Scale. The first two items ask about passive ideation and active ideation, and affirmative responses link to follow-up questions about methods, intent, plans, and attempts. The scale is scored as follows: 0 = no to passive ideation and no to active ideation; 1 = yes to passive ideation (but no to active ideation); 2 = yes to active ideation (but no method, intent, plan); 3 = yes to method (but no intent or plan); 4 = yes to intent (but no plan); 5 = yes to plan; Attempts can be scored on its own or added to the overall scale for a risk score of 6 if participant has a recent suicide attempt.

SECONDARY OUTCOMES:
Youth Risk Behavior Survey Substance Use Questions | Change between baseline and post-intervention/follow-up (12 weeks)
  Measures individual's usage of various substances in their lifetime and within the past 30 days as well as the ways in which individuals have used marijuana, tobacco, or nicotine in the past 30 days. Each substance is individually analyzed for both lifetime usage and past 30 day usage. Individuals can answer Yes or No for both lifetime usage and past 30 day usage. Each substance can range from 0 to the maximum number of survey responses. In addition, for marijuana, students can specify the way in which they used it with response options of smoking, vaping, edible or beverage form, or other. For nicotine and tobacco, students can specify the way in which they used it with the response options of smoking, vaping, or other. "Yes" responses indicate a worse outcome indicating that individuals have used or are currently using the substance in question.
California Healthy Kids Survey General Bullying and Gender Identity/Sexual Orientation-Based Harassment Module | Change between baseline and post-intervention/follow-up (12 weeks)
  Assesses students' perceptions of harassment experiences on school campus among the general student population in addition to bullying and harassment experiences on school campus specific of students who identify as, or are perceived to be, lesbian, gay, bisexual, transgender, questioning, or gender nonconforming.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Goldbach, PhD, Principal Investigator — Washington University School of Medicine
Locations (21):
- United States (21):
  - El Monte High School, El Monte, California
  - Arroyo High School, El Monte, California
  - Fernando R Ledesma High School, El Monte, California
  - Mountain View High School, El Monte, California
  - South El Monte High School, El Monte, California
  - Anderson W. Clark Magnet High School, Glendale, California
  - Animo Leadership High School, Inglewood, California
  - Crescenta Valley High School, La Crescenta-Montrose, California
  - Millikan High School, Long Beach, California
  - Animo Pat Brown Charter High School, Los Angeles, California
  - USC Hybrid High School, Los Angeles, California
  - South LA College Prep, Los Angeles, California
  - Larchmont Charter School, Los Angeles, California
  - Brio College Prep, Los Angeles, California
  - Lynwood High School, Lynwood, California
  - Marco Antonio Firebaugh High School, Lynwood, California
  - Vista High School, Lynwood, California
  - Marshall Fundamental Secondary School, Pasadena, California
  - Blair High School, Pasadena, California
  - Pasadena High School, Pasadena, California
  - Rosemead High School, Rosemead, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT05541406/Prot_002.pdf
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT05541406/ICF_003.pdf